CLINICAL TRIAL: NCT03965715
Title: Development of Energy-storable Ankle-foot Orthosis Using 3D Printing Technology
Brief Title: An Ankle-foot Orthosis Improves Gait Performance and Satisfaction in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A-BR-106-005
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-04

CONDITIONS: Gait Analysis
Keywords: 3D printed technology; Ankle-Foot Orthosis (AFO); Stroke; Gait parameters; Gait Analysis; kinetics; kinematics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gait analysis with barefoot (No Intervention): Participants walk without assistance under gait detection.
- Gait analysis with AFOs (Experimental): Participants walk with AFOs under gait detection.
  Interventions: Device: 3D printing AFO, anterior AFO, off-the-shelf AFO
- Satisfaction questionnaire (Experimental): User feedback from the participants was obtained by questionnaire, the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) and SF-36, to compare the satisfaction of AFOs
  Interventions: Device: 3D printing AFO, anterior AFO, off-the-shelf AFO

INTERVENTIONS:
Device: 3D printing AFO, anterior AFO, off-the-shelf AFO — Subjects wear different AFOs and performed gait analysis.
  Arms: Gait analysis with AFOs; Satisfaction questionnaire

SUMMARY:
All participants were at least 6-month post-stroke and had unilateral limb involvement (8 right/4 left). The main inclusion criteria in selection of the participants in this study were as follows :(1) First stroke (2) At least 6 months post stroke (3) Able to stand for at least one minute without any assistive devices (4) Able to walk for at least 10 meters. All participants were instructed to walk with bare foot or with ankle-foot orthoses(AFOs) separately under gait detection of the motion capture system. Participants were further instructed to complete the 10 Meter Walk Test at a comfortable speed with BF or with AFOs separately. All participants were provided with sufficient rest between each trial. Patient demographics such as lower limb Brunnstrom stage and Modified Ashworth Scale (MAS) score were examined and recorded by experienced therapist. The satisfaction and outcome were measured by the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) and SF-36. The kinematic and kinetic data were collected by Motion Analysis system.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* At least 6 months post-stroke
* Able to stand for at least one minute without any assistive devices
* Able to walk for at least 10 meters.

Exclusion Criteria:

* Unable to walk for at least 10 meters.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-05-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Kinematic analysis | Baseline
  A total of 22 reflective markers were attached to the anatomical landmarks of participants, and a motion capture system with eight cameras was used to collect the kinematics data.
10 Meter Walk Test (10MWT) | Baseline
  Each participant preformed three 10MWT trials under each condition, for a total of 9 trials, on the same day with sufficient time given to rest in between trials.
Numerical rating scale | Baseline
  Participant fatigue before and after the 10MWT for the 3 experimental conditions was measured via a 5-point numerical rating scale (NRS), with 1 indicating no fatigue and 5 indicating strong fatigue.
The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | Baseline
  The 8 items of the questionnaire included Dimensions, Weight, Ease in Adjusting, Safety and Security, Durability , Ease of Use, Comfortable, and Effectiveness. Each item employed a 5-point scale, with 1-point representing not satisfied at all, and 5-point representing very satisfied.
36-Item Short Form Survey (SF-36) | one month after intervention
  The eight-section questionnaire including vitality,physical functioning,bodily pain,general health perceptions, physical role functioning,emotional role functioning,social role functioning,mental health were surveyed to evaluate participant's quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan